CLINICAL TRIAL: NCT01470989
Title: An Open-label Extension Study of CACZ885H2356E2 and CACZ885H2357E2 on the Treatment and Prevention of Gout Flares in Patients With Frequent Flares for Whom NSAIDs and/or Colchicine Are Contraindicated, Not Tolerated or Ineffective
Brief Title: β-RELIEVED - REsponse in Acute fLare and In prEVEntion of episoDes of Re-flare in Gout - Extension 3 (E3)
Acronym: β-RELIEVED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885H2357E3; 2011-003414-17
Record Dates: First submitted 2011-08-16; First posted 2011-11-11 (Estimated); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Acute Gouty Arthritis Flares
Keywords: gouty arthritis
MeSH Terms: conditions — Arthritis, Gouty | interventions — canakinumab; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- canakinumab (Experimental): canakinumab 150 mg s.c.
  Interventions: Drug: ACZ885; Drug: Triamcinolone acetonide 40 mg

INTERVENTIONS:
Drug: ACZ885 — canakinumab 150 mg s.c., given on demand upon new flares
  Other Names: Canakinumab
Drug: Triamcinolone acetonide 40 mg — Participants received 40 mg intramuscular (IM)
  Other Names: Triamcinolone acetonide

SUMMARY:
This was an 18-month, multi-center, open-label, clinical extension study. Patients completing earlier second extension studies (CACZ885H2356E2 and CACZ885H2357E2) continued to be treated in this combined extension 3 study for any new gouty arthritis flare on demand with one subcutaneous (s.c.) injection of canakinumab 150 mg.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed the second extension studies CACZ885H2356E2 or CACZ885H2357E2
* Patients treated with canakinumab in the core studies or subsequent extensions

Exclusion Criteria:

- Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (50):
- United States (31):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Norwalk, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Tustin, California
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Jupiter, Florida
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Wichita, Kansas
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Opelousas, Louisiana
  - Novartis Investigative Site, Flint, Michigan
  - Novartis Investigative Site, Troy, Michigan
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Freehold, New Jersey
  - Novartis Investigative Site, Hickory, North Carolina
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Willoughby Hills, Ohio
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Varnville, South Carolina
  - Novartis Investigative Site, Bristol, Tennessee
  - Novartis Investigative Site, Clarksville, Tennessee
  - Novartis Investigative Site, Johnson City, Tennessee
  - Novartis Investigative Site, Danville, Virginia
  - Novartis Investigative Site, Newport News, Virginia
- Novartis Investigative Site, Darlinghurst, New South Wales, Australia
- Canada (2):
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Novartis Investigative Site, Tallinn, Estonia
- Germany (3):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Magdeburg
- Novartis Investigative Site, Valmiera, Latvia
- Lithuania (4):
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Šiauliai
  - Novartis Investigative Site, Vilnius
- Russia (5):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Ukraine (2):
  - Novartis Investigative Site, Uzhhorod
  - Novartis Investigative Site, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 60 centers from 10-November-2011 (first participant first visit) to 22-May-2013 (last participant last visit).
Pre-assignment Details: A total of 456 participants were randomized in the core studies (CACZ885H2356 and CACZ885H2357) of which 335 participants entered the first extension (CACZ885H2356E2) study. Out of the 317 participants who completed the first extension studies, 272 participants entered the second extension studies(CACZ885H2357E2 ). Out of the 249 participants who completed the second extension studies 136 participants entered the third extension study(CACZ885H2357E3).
Groups:
- Canakinumab 150 mg: Participants received 150 mg subcutaneously (S.C) at randomization and upon new flare. The doses were provided as pre-filled syringes.
- Triamcinolone Acetonide 40 mg: Participants received 40 mg intramuscular (IM) at randomization and upon new flare.
Period: Overall Study
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Started | 227 | 229
Completed Core Study | 208 | 208
Entered Extension 1 Study | 174 | 161
Completed Extension 1 Study | 165 | 152
Entered Extension 2 Study | 141 | 131
Completed Extension 2 Study | 132 | 117
Entered Extension 3 | 87 | 49
Completed | 79 | 43
Not Completed | 148 | 186
Not completed — Participants did not entered extension studies 1, 2 and 3 | 103 | 136
Not completed — Adverse Event | 2 | 5
Not completed — Abnormal laboratory value | 1 | 1
Not completed — Unsatisfactory therapeutic effect | 0 | 6
Not completed — Withdrawal by Subject | 19 | 17
Not completed — Lost to Follow-up | 18 | 13
Not completed — Administrative problems | 2 | 4
Not completed — Death | 2 | 2
Not completed — Protocol deviation | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Set consists of all participants that received study drug in the core study and had at least one post-baseline safety assessment.
  The demographic data was not combined for the E3 analysis.
Groups:
- Triamcinolone Acetonide 40 mg: Participants received 40 mg Triamcinolone Acetonide intramuscular (IM) at randomization and upon new flare and re-treated with at least 1 dose of canakinumab.
- Total: Total of all reporting groups
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg | Total
Number analyzed (Participants) | 225 | 229 | 454
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The mean value given here is from the CACZ885H2356E2 study.
  years
    number analyzed (Participants) | 113 | 115 | 228
    (all) | 54.0 (11.8) | 54.6 (10.71) | 54.3 (10.93)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The mean value given here is from the CACZ885H2357E2 study.
  years
    number analyzed (Participants) | 112 | 114 | 226
    (all) | 50.6 (12.10) | 52.6 (12.28) | 51.6 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The value given here is from the CACZ885H2356E2 study.
  Participants
    number analyzed (Participants) | 113 | 115 | 228
    Female | 12 | 7 | 19
    Male | 101 | 108 | 209
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The value given here is from the CACZ885H2357E2 study.
  Participants
    number analyzed (Participants) | 112 | 114 | 226
    Female | 12 | 9 | 21
    Male | 100 | 105 | 205
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The value given here is from the CACZ885H2356E2 study.
  Participants
    Caucasian: number analyzed (Participants) | 113 | 115 | 228
    Caucasian | 93 | 96 | 189
    Asian: number analyzed (Participants) | 113 | 115 | 228
    Asian | 3 | 3 | 6
    Native American: number analyzed (Participants) | 113 | 115 | 228
    Native American | 1 | 1 | 2
    Other: number analyzed (Participants) | 113 | 115 | 228
    Other | 16 | 15 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The value given here is from the CACZ885H2357E2 study.
  Participants
    Caucasian: number analyzed (Participants) | 112 | 114 | 226
    Caucasian | 74 | 80 | 154
    Black: number analyzed (Participants) | 112 | 114 | 226
    Black | 26 | 24 | 50
    Asian: number analyzed (Participants) | 112 | 114 | 226
    Asian | 10 | 9 | 19
    Other: number analyzed (Participants) | 112 | 114 | 226
    Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Incidence Rate (IR) of Adverse Events, Serious Adverse Events and Death Per 100 Patient-years in Participants
Description: Adverse events (AEs) were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline,or, if present at baseline, appears to worsen. Serious adverse events (SAEs) were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards.
Time Frame: From start of the core studies (CACZ885H2357 [NCT01080131] and CACZ885H2361 [NCT01356602]) up to end of the current study (36 weeks)
Population: The Safety Set consists of all participants that received study drug in the core study and had at least one post-baseline safety assessment.
Measure: Number; unit: IR/100 patient-years
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 225 | 229
IR/100 patient-years
  Adverse Events | 873 | 451
  Non Fatal SAEs | 59 | 25
  Death | 2 | 2

2. Secondary Outcome: Number of New Flares Per Participant
Description: Flare rate was calculated as the number of new flares over the period of observation in years. New flares occurred before first study medication dose in extension 3 study were considered.
Time Frame: as for outcome 1
Population: Modified Analysis Set (MAS) consisted of all participants randomized in the core studies and received both treatments according to their exposure.
Measure: Mean (Standard Deviation); unit: flares
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
Number analyzed (Participants) | 225 | 229
flares | 1.109 (1.608) | 2.459 (3.701)

3. Secondary Outcome: Patient's Assessment of Gout Pain Intensity in the Most Affected Joint
Description: Participant scored their current pain intensity in the most affected joint of the gout flare on a 5-point Likert Scale (none or mild).
Time Frame: up to 7 days post-dose
Population: Modified Analysis Set (MAS) consisted of all Full Analysis Set (FAS) participants. The FAS consisted of all enrolled participants who have received at least one dose of study medication. This outcome measure was assessed only in the subset of participants who had re-treatment with at least one dose of canakinumab.
Measure: Count of Participants; unit: Participants
Groups:
- Canakinumab Retreatment: Participants received 150 mg canakinumab subcutaneously (S.C) at randomization and upon new flare and re-treated with at least 1 dose of canakinumab.
- Triamcinolone Acetonide- Randomized to Canakinumab Treatment: Participants received 40 mg Triamcinolone Acetonide intramuscular (IM) at randomization and upon new flare and re-treated with at least 1 dose of canakinumab.
Arm/Group | Canakinumab Retreatment | Triamcinolone Acetonide- Randomized to Canakinumab Treatment
Number analyzed (Participants) | 127 | 78
Participants
  Baseline Flare | 102 | 72
  Last New Flare | 104 | 69

ADVERSE EVENTS:
Time Frame: Adverse Event were Collected From start of the core studies (CACZ885H2357 [NCT01080131] and CACZ885H2361 [NCT01356602]) up to end of the current study (36 weeks)
Description: The Safety Set consists of all participants that received study drug in the core study and had at least one post-baseline safety assessment.
Arm/Group | Canakinumab 150 mg | Triamcinolone Acetonide 40 mg
All-Cause Mortality (participants affected / at risk) | 2/225 | 2/229
Serious Adverse Events (participants affected / at risk) | 35/225 | 23/229
Other Adverse Events (participants affected / at risk) | 87/225 | 55/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab 150 mg (N=225) | Triamcinolone Acetonide 40 mg (N=229)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 2
Angina unstable (Cardiac disorders) | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Periproctitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Cyst (General disorders) | 1 | 0
Device dislocation (General disorders) | 1 | 0
Hernia obstructive (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Abscess jaw (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Prostatic specific antigen increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 0
Convulsion (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 2
Spinal cord ischaemia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Vesical fistula (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab 150 mg (N=225) | Triamcinolone Acetonide 40 mg (N=229)
Nasopharyngitis (Infections and infestations) | 8 | 12
Upper respiratory tract infection (Infections and infestations) | 18 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 | 6
Headache (Nervous system disorders) | 14 | 10
Hypertension (Vascular disorders) | 29 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No